CLINICAL TRIAL: NCT00710203
Title: Efficacy of a 585 nm Pulsed Dye Laser (PDL) for the Treatment of Dermatosis Papulosa Nigra, and Compare it to Therapy With Curettage and Electrodesiccation.
Brief Title: Dermatosis Papulosa Nigra
Acronym: DPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 200715981
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Facial Dermatoses; Seborrheic Keratoses
Keywords: Dermatosis Papulosa Nigra; seborrheic keratoses
MeSH Terms: conditions — Facial Dermatoses; Keratosis, Seborrheic; Dermatosis Papulosa Nigra | interventions — Lasers, Dye; Curettage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pulsed dye laser (Active Comparator): Four lesions are selected on each subject for study. One lesion will be chosen for treatment with the pulsed dye laser with a 7 mm spot size. A single 10 J/cm2 pulse with 10 ms pulse duration will be used to treat the lesion.
  Interventions: Device: Pulsed dye laser
- Curettage (Active Comparator): Four lesions are selected on each subject for study. A second lesion will be treated with curettage with or without anesthetic, depending on the patient's preference.
  Interventions: Procedure: Curettage
- Electrodesiccation (Active Comparator): Four lesions are selected on each subject for study. A third lesion will be treated with electrodesiccation after infiltration of 1% lidocaine with epinephrine.
  Interventions: Procedure: Electrodesiccation
- No treatment (Active Comparator): Four lesions are selected on each subject for study. A fourth lesion will not be treated and will serve as a control.
  Interventions: Other: No treatment

INTERVENTIONS:
Device: Pulsed dye laser — One lesion will be chosen for treatment with the pulsed dye laser with a 7 mm spot size. A single 10 J/cm2 pulse with 10 ms pulse duration will be used to treat the lesion.
  Other Names: The study will involve the use of Cynosure Cynergy 585 nm Pulsed Dye LASER.
  Arms: Pulsed dye laser
Procedure: Curettage — A second lesion will be treated with curettage with or without anesthetic, depending on the patient's preference.
  Arms: Curettage
Procedure: Electrodesiccation — A third lesion will be treated with electrodesiccation after infiltration of 1% lidocaine with epinephrine.
  Arms: Electrodesiccation
Other: No treatment — A fourth lesion will not be treated and will serve as a control.
  Arms: No treatment

SUMMARY:
DPN is a disorder among darkly pigmented patients, manifested by small, benign, variants of seborrheic keratoses, predominantly on the face.

The purpose of this study is to determine the efficacy of a 585 nm PDL for the treatment of Dermatosis Papulosa Nigra, and compare it to therapy with curettage (scraping the lesions off) and electrodesiccation (burning the lesions off).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Able to give informed consent.
* Desires removal of lesions.
* Willing to come back for six week follow-up.
* Willing to fill out post operative questionnaire.
* At least 4 lesions less than 7 mm.
* Diagnosis of Dermatosis Papulosa Nigra (DPN)

Exclusion Criteria:

* Less than 18 years of age.
* Pregnant.
* Sensitive to laser energy.
* History of Collagen Vascular Disorders.
* History of Keloids.
* History of post inflammatory hyperpigmentation.
* Incarcerated.
* Unable to give informed consent.
* Unable to follow up for post operative evaluation.
* Unable to complete patient visual analogue scale.
* Unable to understand consent process or risks.
* Unable to accept risk of scar, infection, minor bleeding, permanent or prolonged hyperpigmentation and hypopigmentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm: 10 patients will be recruited from the University of California, Davis Department of Dermatology. Digital images will be taken immediately prior to treatment. One lesion will be chosen for treatment with the pulsed dye laser with a 7 mm spot size. A single 10 J/cm2 pulse with 10 ms pulse duration will be used to treat the lesion. A second lesion will be treated with curettage with or without anesthetic, depending on the patient's preference, and a third lesion will be treated with electrodesiccation after infiltration of 1% lidocaine with epinephrine. A fourth lesion will not be treated and will serve as a control.
Period: Overall Study
Arm/Group | Study Arm
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.60 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Clearance of All Lesions
Description: The physician assessed percent clearance of all treated lesions and the control lesion.
Time Frame: 6 to 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of lesion clearance
Units Other Than Participants: lesions
Arm/Group | Pulsed Dye Laser | Curettage | Electrodesiccation | No Treatment
Number analyzed (Participants) | 10 | 10 | 10 | 10
Number analyzed (lesions) | 10 | 10 | 10 | 10
percentage of lesion clearance | 88 (24.06) | 96 (16.87) | 92.5 (9.661) | 0 (0)

2. Other Pre Specified Outcome: Evidence of Hypopigmentation
Description: The physician assessed evidence of hypopigmentation.
Time Frame: 6 to 12 weeks
Measure: Number; unit: lesions
Arm/Group | Pulsed Dye Laser | Curettage | Electrodesiccation | No Treatment
Number analyzed (Participants) | 10 | 10 | 10 | 10
lesions | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Evidence of Hyperpigmentation
Description: The physician assessed evidence of hyperpigmentation.
Time Frame: 6 to 12 weeks
Measure: Number; unit: lesions
Arm/Group | Pulsed Dye Laser | Curettage | Electrodesiccation | No Treatment
Number analyzed (Participants) | 10 | 10 | 10 | 10
lesions | 4 | 4 | 5 | 0

4. Other Pre Specified Outcome: Evidence of Scar
Description: The physician assessed evidence of scar.
Time Frame: 6 to 12 weeks
Measure: Number; unit: lesions
Arm/Group | Pulsed Dye Laser | Curettage | Electrodesiccation | No Treatment
Number analyzed (Participants) | 10 | 10 | 10 | 10
lesions | 0 | 0 | 0 | 0

5. Other Pre Specified Outcome: Evidence of Texture Irregularities
Description: The physician assessed evidence of texture irregularities.
Time Frame: 6 to 12 weeks
Measure: Number; unit: lesions
Arm/Group | Pulsed Dye Laser | Curettage | Electrodesiccation | No Treatment
Number analyzed (Participants) | 10 | 10 | 10 | 10
lesions | 1 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Description: No serious and/or other (non-serious) adverse events were observed.
Groups:
- Pulsed Dye Laser: 10 patients will be recruited from the University of California, Davis Department of Dermatology. Digital images will be taken immediately prior to treatment. Four lesions are selected on each subject for study. One lesion will be chosen for treatment with the pulsed dye laser with a 7 mm spot size. A single 10 J/cm2 pulse with 10 ms pulse duration will be used to treat the lesion.
- Curettage: 10 patients will be recruited from the University of California, Davis Department of Dermatology. Digital images will be taken immediately prior to treatment. Four lesions are selected on each subject for study. A second lesion will be treated with curettage with or without anesthetic, depending on the patient's preference.
- Electrodesiccation: 10 patients will be recruited from the University of California, Davis Department of Dermatology. Digital images will be taken immediately prior to treatment. Four lesions are selected on each subject for study. A third lesion will be treated with electrodesiccation after infiltration of 1% lidocaine with epinephrine.
- No Treatment: 10 patients will be recruited from the University of California, Davis Department of Dermatology. Digital images will be taken immediately prior to treatment. Four lesions are selected on each subject for study. A fourth lesion will not be treated and will serve as a control.
Arm/Group | Pulsed Dye Laser | Curettage | Electrodesiccation | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No